CLINICAL TRIAL: NCT06938828
Title: Physiotherapy in the Treatment of Patients With Neck Pain After a Commuting Accident; a Retrospective Cohort Study
Brief Title: Treatment of Patients With Neck Pain After a Commuting Accident
Status: Active, not recruiting | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, Principal Investigator, Universidad Católica San Antonio de Murcia
Other Study IDs: Itinere
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Cervical Injury Spine
Keywords: neck pain; physiotherapy; accidents in itinere; Incapacity for work
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational group: Data will be collected from medical records of a mutual insurance company that collaborates with the Social Security. The data will be from patients of both sexes with a medical diagnosis of neck pain secondary to traffic accidents while commuting and without a medical diagnosis of associated traffic pathology, between the years 2022 and 2024. The patients had received a physiotherapy intervention with and without manual therapy.
  Interventions: Other: Observational cohort group

INTERVENTIONS:
Other: Observational cohort group — As this is an observational cohort study, there will be no intervention. In this study, only retrospective data will be collected for subsequent analysis. Similarly, the aim is to assess the relationship between the time on sick leave and the type of physiotherapy treatment received by patients. As this is an observational and retrospective cohort study, there is no risk derived from the development of the study for the subjects whose data form part of the study.

SUMMARY:
Introduction. Neck pain is one of the main causes of incapacity for work. The economic impact of neck pain is considerable due to the cost of medical treatment and physiotherapy. Accidents in itinere, those that occur on the way between home and the workplace, can cause pain and functional impairment.

Objective. To analyze the relationship between the time off work following accidents on the way to and from work and the type of treatment received.

Material and method. Multicenter retrospective cohort study. Data will be collected from 146 patients. The primary variable of the study will be the time on sick leave (in days), with the type of intervention received (manual therapy or not) being the dependent variable. The secondary variables, estimated as modifying or confounding, will be the intensity of the pain (visual analog scale), sex, age, occupational cervical strain, type of contract (salaried/self-employed) and the number of physiotherapy sessions received.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Persons aged 18 to 65
* Patients with a medical diagnosis of neck pain secondary to traffic accidents while commuting
* Persons without a medical diagnosis of another associated pathology
* Patients whose accident occurred between 2022 and 2024.

Exclusion Criteria:

* Patients who have received physiotherapy treatment at another centre during the process
* Patients who requested voluntary discharge for whatever reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have suffered a traffic accident while traveling to or from work between 2022 and 2024.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-05-13 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Measurement of time off work | Screening visit
  The dependent variable, time off work, will be measured in days.

SECONDARY OUTCOMES:
Measurement of type of intervention received | Screening visit
  The secondary variable, type of intervention received, will be evaluated with a dichotomous coding: manual therapy or no manual therapy.
Measurement of pain intensity at the time of medical discharge | Screening visit
  The secondary variable, pain intensity at the time of medical discharge, will be collected with the recording of the visual analog scale (range 0-10)
Measurement of the number of physiotherapy sessions received | Screening visit
  The secondary variable, number of physiotherapy sessions received, will be measured quantitatively (in days of treatment administration). This value will be collected from the physiotherapy record
Measurement of the type of employment contract of the patients | Screening visit
  The secondary variable, type of employment contract of the patients, will be collected in a dichotomous qualitative variable (salaried/self-employed)
Measuring the age of the patients | Screening visit
  The secondary variable, age of the patients, will be collected in a quantitative variable of completed years (measured in days)
Measurement of patients' occupational cervical strain | Screening visit
  The secondary variable, patients' cervical strain , will be collected in a qualitative variable (Yes/No) depending on the type of work of the patients, their daily work may or may not require cervical strain.
Measuring the gender of patients | Screening visit
  The secondary variable, the gender of patients, will be collected in a qualitative variable (Female/Male).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica San Antonio de Murcia, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided